CLINICAL TRIAL: NCT04140448
Title: Ultra-wide-field Fluorescein Angiography in Patients With Macular Edema Secondary to Retinal Vein Occlusion
Acronym: UWFA-RVO-ME
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Renmin Hospital of Wuhan University (Other)
Responsible Party: Principal Investigator, Changzheng Chen, Chief of Department of Ophthalmology, Renmin Hospital of Wuhan University
Other Study IDs: UWFA-RVO-ME
Record Dates: First submitted 2019-10-24; First posted 2019-10-25 (Actual); Last update posted 2023-10-18 (Actual); Status verified 2023-10

CONDITIONS: Retinal Vein Occlusion; Macular Edema
Keywords: Ultra-wide field fundus fluorescein angiography; ischemic index; leakage index
MeSH Terms: conditions — Retinal Vein Occlusion; Macular Edema | interventions — Ranibizumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- UWFA-RVO-ME: Ultra-wide-field fundus fluorescein angiography on patients with macular edema secondary to retinal vein occlusion treated with Ranibizumab
  Interventions: Drug: Ranibizumab 0.5 MG/0.05 ML Intraocular Solution [LUCENTIS]; Device: Ultra-wide Fluorescein Angiography

INTERVENTIONS:
Drug: Ranibizumab 0.5 MG/0.05 ML Intraocular Solution [LUCENTIS] — Intravitreal injection of Ranibizumab 0.5 MG/0.05 ML
  Other Names: Lucentis; Anti-VEGF
Device: Ultra-wide Fluorescein Angiography — Ultra-wide-field Fluorescein Angiography can clearly observe the peripheral retina

SUMMARY:
This study mainly observed the ischemic index and vascular leakage index changes on ultra-wide field fluorescence angiography after anti-VEGF treatment , and whether these changes correlated with treatment efficacy in patients with macular edema secondary to retinal vein occlusion.

DETAILED DESCRIPTION:
Ultra-wide field fluorescence angiography can clearly observe the peripheral retina. This study mainly observes the ischemic index and vascular leakage index changes on UWFA after anti-VEGF treatment and evaluates these changes associated with treatment efficacy in patients with macular edema secondary to retinal vein occlusion.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female aged 18 years or older
2. Macular edema secondary to CRVO,BRVO or HRVO
3. Duration of RVO not more than 4 months
4. Naïve patients. Patient with previous RVO (more than 12 months before the inclusion date) completely resolved (normalization of visual acuity and fundus examination) and who have experienced a recurrence of RVO are also considered naive
5. Patient who agrees to participate in the study and who has given his/her written, informed consent

Exclusion Criteria:

1. Patient with another retinal disease in the study eye: diabetic retinopathy, maculopathy of any cause (age-related macular degeneration, epimacular membrane, myopia, etc) responsible for decreased vision, advanced glaucoma, cataract severely affecting vision and/or requiring surgical treatment during the 24 months study period
2. Active or suspected ocular or periocular infection
3. Active severe intraocular inflammation
4. RVO complicated with neovascularization
5. Patient who has previously undergone laser panretinal photocoagulation, grid-laser or photodynamic therapy, any anti-VEGF or corticoids intravitreal injections in the study eye
6. Patient already included in the study for the treatment of the fellow eye
7. Pregnant or breastfeeding woman
8. Lack of effective contraception for women of childbearing age
9. Patient taking part in an interventional study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Chinese
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2023-10-09 (Estimated); Primary Completion 2024-10-30 (Estimated); Study Completion 2025-12-15 (Estimated)

PRIMARY OUTCOMES:
Change in vascular leakage index in different retinal area | Baseline and 1,2,3,4,6,9 and 12 months
  Change in vascular leakage index in different retinal area from baseline to 1,2,3,4,6,9 and 12 months
Change in non-perfused areas in different retinal area | Baseline and 1,2,3,4,6,9 and 12 months
  Change in non-perfused areas in different retinal area from baseline to 1,2,3,4,6,9 and 12 months

SECONDARY OUTCOMES:
Change in best corrected visual acuity | Baseline and 1,2,3,4,6,9 and 12 months
  Change in best corrected visual acuity from baseline to 1,2,3,4,6,9 and 12 months
Change in central macular thickness | Baseline and 1,2,3,4,6,9 and 12 months
  Change in central macular thickness from baseline to1,2,3,4,6,9 and12 months

CONTACTS AND LOCATIONS:
Overall Officials: CZ Chen, PHD, Principal Investigator — Renmin Hospital of Wuhan University
Locations (1):
- Renmin Hospital of Wuhan University, Wuhan, Hubei, China